CLINICAL TRIAL: NCT03216382
Title: The Impact of the Attention Training Technique on Attention Control and High Worry
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Toronto Metropolitan University (Other)
Collaborators: Ministry of Research, Innovation and Science, Ontario (Other)
Responsible Party: Principal Investigator, Kathleen Stewart, Graduate Student, Toronto Metropolitan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017-186
Record Dates: First submitted 2017-07-11; First posted 2017-07-13 (Actual); Results first posted 2021-07-02 (Actual); Last update posted 2021-07-02 (Actual); Status verified 2021-06

CONDITIONS: Excessive Worry
Keywords: High worry; Anxiety; Attention Training Technique; Attention Control; Attention; Mindfulness; Attention Bias; Worry; Pathological Worry; Anxiety Disorder
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Baseline outcome measures will be completed at the first visit to the lab. Participants will then engage in a week of reporting on their worry and attention on their own, before coming back to the lab to recomplete the outcome measures. They will then be randomly assigned to the intervention or control condition and will engage in a week of daily listening to the corresponding recording for their condition on their own, while reporting on their worry and attention again during that week. Outcome measures will be completed again at the lab immediately following the intervention.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Attention Training Technique (Experimental): Participants in this arm will listen to the Attention Training Technique. Participants will listen to the recording once in the lab, followed by a week of once/day listening at home for a week. For a week before the intervention, and for the week during the intervention, participants will respond to questions every evening, about their worry and attention that day.
  Interventions: Behavioral: Attention Training Technique
- Control Condition (Placebo Comparator): Participants in this arm will listen to the control condition recording. Participants will listen to the recording once in the lab, followed by a week of once/day listening at home for a week. For a week before the intervention, and for the week during the intervention, participants will respond to questions every evening, about their worry and attention that day.
  Interventions: Behavioral: Control Condition

INTERVENTIONS:
Behavioral: Attention Training Technique — The ATT is a 12-minute audio recording that includes sounds and a voice guiding attention to the sounds. The sounds play continuously during the training task.
  Arms: Attention Training Technique
Behavioral: Control Condition — In the control condition, participants listen to an audio recording with the same sounds as the ATT recording, and a voice that delivers placebo instructions.
  Arms: Control Condition

SUMMARY:
Excessive and uncontrollable worry has been associated with deficits in attention control. The Attention Training Technique (ATT; Wells, 1990) is a 12-minute audio recording that was developed to train attention control, so that individuals could learn to shift their attention away from maladaptive cognitive processes such as worry. The technique has shown to be promising at reducing symptoms across a variety of mental disorders (Knowles, Foden, El-Deredy, & Wells, 2016) and is recommended for use in people who suffer from chronic worry. To date, little research has been conducted examining the benefits of using this technique in such a population. The present study aims to examine the immediate and short term effects of weekly ATT practice, compared to a control condition, in a population that suffers from high levels of worry about a variety of topics. About one-hundred participants who suffer from chronic worry will be randomly assigned to listen to the ATT or a control recording, every day for a week. Changes in attention control, worry, and cognitive processes will be examined over the course of the intervention period.

DETAILED DESCRIPTION:
People who suffer from pathological worry report that they worry to an excessive degree and that they find it very difficult to control their worry. Deficits in attention control may help to explain why people who worry pathologically find it difficult to shift their attention away from their worry, and back to the task at hand. The Attention Training Technique (ATT; Wells, 1990) was developed to train attentional control, so that individuals could learn to shift the focus of their attention away from maladaptive cognitive processes such as worry. Despite being recommended for use in populations that suffer from excessive worry, there is a dearth of research examining the effects of ATT in such a population. The study aims to examine the immediate (during the intervention) and short-term (right after finishing the intervention) effects of listening to the ATT, compared to the control recording, on attention, worry, and other cognitive processes. This will be the first study to our knowledge to examine the effects of 1 week of daily ATT practice in a sample of people who suffer from chronic worry, and will provide important information for optimizing the treatment of worry in this population.

ELIGIBILITY:
Inclusion Criteria:

1. Score of 65 or higher on the Penn State Worry Questionnaire.
2. Endorsement of chronic worry as per the description of Generalized Anxiety Disorder (GAD) (American Psychiatric Association, 2013).

Exclusion Criteria:

1. Has current or past history of psychosis or mania, or endorse symptoms consistent with a diagnosis of a substance use disorder in the past 12 months
2. Report clinically significant suicidal ideation, intent, or plan
3. Participants will be excluded if they are currently receiving psychological treatment or counseling (e.g., cognitive behaviour therapy, supportive counseling, etc.), unless this treatment is infrequent (once monthly or less) or the participant has been receiving consistent weekly treatment for at least 12 weeks and still meets all other eligibility criteria
4. Are taking psychotropic medications and have had a change in dose in the past 12 weeks. If they have recently discontinued a psychotropic medication, they will be included if it has been at least 1 month since discontinuation, or 3 months if they had been taking fluoxetine/Prozac. If a participant is taking benzodiazepines on an 'as needed' basis they will be included and their use of this medication will be noted. Daily benzodiazepine usage will exclude participants, and if participants have ever taken benzodiazepines daily, they must be abstinent for at least one year.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2017-08-15 (Actual); Primary Completion 2019-06-26 (Actual); Study Completion 2019-06-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen E Stewart, Bsc, Principal Investigator — Toronto Metropolitan University
Locations (1):
- Ryerson University, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Results of the study will be disseminated via conference presentations, journal publications, and through our lab website. Upon request, de-identified aggregate participant data may be made available to a publishing journal or individual research group. Individual research groups interested in accessing de-identified data will be required to submit a proposal detailing their intended use of the data. Their qualifications will be reviewed based on their proposal and CVs. Individual research groups approved for access will be required to agree to not attempt to re-identify participants, not further distribute data, and not use the data for purposes other than specified in their original proposal. No individual data will be shared.

REFERENCES:
- [Background] Wells A. Panic disorder in association with relaxation induced anxiety: An attentional training approach to treatment. Behavior Therapy, 21(3): 273-280, 1990.
- [Background] Knowles MM, Foden P, El-Deredy W, Wells A. A Systematic Review of Efficacy of the Attention Training Technique in Clinical and Nonclinical Samples. J Clin Psychol. 2016 Oct;72(10):999-1025. doi: 10.1002/jclp.22312. Epub 2016 Apr 29. PMID 27129094
- [Derived] Stewart KE, Antony MM, Koerner N. A randomized experimental analysis of the attention training technique: Effects on worry and relevant processes in individuals with probable generalized anxiety disorder. Behav Res Ther. 2021 Jun;141:103863. doi: 10.1016/j.brat.2021.103863. Epub 2021 Apr 10. PMID 33872957
- See also: Lab Website — http://psychlabs.ryerson.ca/caplab/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited with flyers and online advertisements. Recruitment took place between 2017-2019 at Ryerson University, Toronto, Ontario, Canada.
Period: Overall Study
Arm/Group | Attention Training Technique | Control Condition
Started | 41 | 54
Completed | 34 | 44
Not Completed | 7 | 10

BASELINE CHARACTERISTICS:
Population: Complete case analysis was used, thus only participants who completed the entire intervention were included in the baseline analyses.
Groups:
- Total: Total of all reporting groups
Arm/Group | Attention Training Technique | Control Condition | Total
Number analyzed (Participants) | 34 | 44 | 78
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 34 | 44 | 78
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.15 (12.35) | 23.89 (11.25) | 29.44 (11.68)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender: Female | 26 | 38 | 64
  Gender: Male | 8 | 5 | 13
  Gender: Other | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: White | 12 | 11 | 23
  Ethnicity: Southeast Asian | 5 | 13 | 18
  Ethnicity: South Asian | 5 | 7 | 12
  Ethnicity: East Asian | 3 | 8 | 11
  Ethnicity: Latin American | 3 | 0 | 3
  Ethnicity: Mixed | 3 | 2 | 5
  Ethnicity: Black | 2 | 1 | 3
  Ethnicity: Arab/West Asian | 1 | 0 | 1
  Ethnicity: Other | 0 | 1 | 1
  Ethnicity: Aboriginal | 0 | 1 | 1
Penn State Worry Questionnaire [Mean (Standard Deviation); unit: units on a scale] — Range: 16-80 Greater scores indicate greater pathological worry
  units on a scale | 70.18 (4.08) | 70.79 (3.69) | 70.53 (3.85)
Generalized Anxiety Disorder Questionnaire-IV [Mean (Standard Deviation); unit: units on a scale] — Range: 0-12 Greater scores include greater GAD symptom severity
  units on a scale | 10.39 (1.89) | 10.04 (2.20) | 10.19 (2.06)
Center for Epidemiologic Studies Depression Scale-Revised [Mean (Standard Deviation); unit: units on a scale] — Range: 0- 60 Greater scores represent greater depression symptom severity
  units on a scale | 27.53 (13.25) | 28.25 (12.96) | 27.94 (13.01)

OUTCOME MEASURES:

1. Primary Outcome: Breathing Focus Task -Negative Intrusions
Description: Behavioural measure of attention control over worry. Number of negative thought intrusions reported during the post-worry breathing focus period (i.e. a period of focused breathing after a period of worry). Scores range from 0-12. A greater number means more negative thought intrusions.
Time Frame: Administered three times over the course of two weeks. Changes will be examined from Visit 1 (Baseline) to Visit 2 (Preintervention, 1 week following Baseline) and Visit 2 to Visit 3 (1 week following preintervention).
Population: Participants were only included on this analyses if they had data for all time points. 3 participants were not included (1 from ATT, 2 from control).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Attention Training Technique | Control Condition
Number analyzed (Participants) | 33 | 42
score on a scale
  Visit 1 | 2.85 (2.32) | 2.55 (1.99)
  Visit 2 | 2.45 (2.53) | 2.26 (1.93)
  Visit 3 | 1.79 (2.13) | 1.64 (1.82)
Statistical Analysis 1: Comparison: Attention Training Technique vs Control Condition; Test type: Superiority; p = .93, ANOVA — The apriori threshold for significance was a = 0.05. The p value reflects the test of an interaction between condition and time

2. Primary Outcome: Daily Worry Questions
Description: A daily self-report measure of the frequency, duration, intensity and uncontrollability of worry. Only uncontrollability of worry was used (see Data Analysis Plan for rationale). Scores range from 0-6. Higher scores represent greater uncontrollability of worry.
Time Frame: Completed every evening for two weeks. The first week will take place before beginning the ATT/ control intervention. The second week will take place during the intervention period.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Attention Training Technique | Control Condition
Number analyzed (Participants) | 34 | 44
units on a scale
  Day 1 | 3.66 (1.14) | 3.15 (1.52)
  Day 2 | 3.56 (1.83) | 3.63 (1.70)
  Day 3 | 2.86 (1.78) | 3.34 (1.83)
  Day 4 | 3.48 (1.75) | 3.28 (1.80)
  Day 5 | 3.34 (1.50) | 3.41 (1.62)
  Day 6 | 3.11 (1.50) | 3.17 (1.54)
  Day 7 | 3.56 (1.48) | 3.18 (1.66)
  Day 8 | 3.55 (1.60) | 3.56 (1.52)
  Day 9 | 2.87 (1.52) | 3.43 (1.69)
  Day 10 | 3.13 (1.79) | 3.63 (1.54)
  Day 11 | 3.28 (1.45) | 3.13 (1.53)
  Day 12 | 3.15 (1.78) | 3.44 (1.98)
  Day 13 | 3.31 (1.61) | 3.11 (1.67)
  Day 14 | 2.97 (1.54) | 3.03 (1.67)
Statistical Analysis 1: Comparison: Attention Training Technique vs Control Condition; HLM piecewise analysis was used to examine linear change from day 1-7 (visit 1 to visit 2) and change from day 7-14 (visit 2 to visit 3) on uncontrollability of worry; Test type: Superiority; p = .74, Mixed Models Analysis — this value represents the interaction between condition and the intervention time period The apriori threshold for significance was a = 0.05
Statistical Analysis 2: Comparison: Attention Training Technique vs Control Condition; HLM piecewise analysis was used to examine quadratic change from day 1-7 (visit 1 to visit 2) and change from day 7-14 (visit 2 to visit 3) on uncontrollability of worry; Test type: Superiority; p = .44, Mixed Models Analysis — this value represents the interaction between condition and the intervention time period (squared) The apriori threshold for significance was a = 0.05

3. Secondary Outcome: Penn State Worry Questionnaire-Past Week
Description: Self-report measure of the degree of worry experienced over the past week. Scores range from 15 to 75. Higher scores indicate higher worry over the past week.
Time Frame: as for outcome 1
Population: Participants were only included on this analyses if they had data for all time points. 1 participant was not included from the control condition.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Attention Training Technique | Control Condition
Number analyzed (Participants) | 34 | 43
score on a scale
  Visit 1 | 71.91 (9.23) | 72.72 (8.69)
  Visit 2 | 67.38 (13.15) | 67.51 (12.13)
  Visit 3 | 61.06 (13.51) | 63.07 (15.41)
Statistical Analysis 1: Comparison: Attention Training Technique vs Control Condition; Test type: Superiority; p = .17, ANOVA — the apriori threshold for significance was a = 0.05 The p value reflects the test of an interaction between condition and time

4. Secondary Outcome: Self-Attention Rating Scale
Description: A daily self-report measure of focus of attention (from internal to externally focused). The scale ranges from 0 to 6. 0 represents entirely externally focused and 6 represents entirely internally focused.
Time Frame: Completed before and after listening to the recoding (immediate change) and every evening for two weeks. The first week will take place before beginning the ATT/ control intervention. The second week will take place during the intervention period.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Attention Training Technique | Control Condition
Number analyzed (Participants) | 33 | 44
units on a scale
  Day 1 | 3.72 (1.41) | 3.56 (1.37)
  Day 2 | 3.11 (1.67) | 3.11 (1.56)
  Day 3 | 3.18 (1.49) | 3.69 (1.51)
  Day 4 | 3.17 (1.50) | 3.00 (1.58)
  Day 5 | 3.61 (1.40) | 3.00 (1.76)
  Day 6 | 3.75 (1.62) | 3.64 (1.66)
  Day 7 | 4.11 (1.50) | 3.33 (1.69)
  Day 8 | 3.03 (1.30) | 3.44 (1.50)
  Day 9 | 2.87 (1.71) | 3.30 (1.33)
  Day 10 | 3.48 (1.88) | 3.25 (1.55)
  Day 11 | 3.06 (1.59) | 3.29 (1.45)
  Day 12 | 3.08 (1.79) | 3.27 (1.50)
  Day 13 | 3.41 (1.59) | 3.18 (1.41)
  Day 14 | 3.69 (1.42) | 3.05 (1.63)
Statistical Analysis 1: Comparison: Attention Training Technique vs Control Condition; HLM piecewise analysis was used to examine linear change from day 1-7 (visit 1 to visit 2) and change from day 7-14 (visit 2 to visit 3) on self-focused attention; Test type: Superiority; p = .50, Mixed Models Analysis — The apriori threshold for significance was a = 0.05 The p value reflects the test of an interaction between condition and time
Statistical Analysis 2: Comparison: Attention Training Technique vs Control Condition; HLM piecewise analysis was used to examine quadratic change from day 1-7 (visit 1 to visit 2) and change from day 7-14 (visit 2 to visit 3) on self-focused attention; Test type: Superiority; p = .02, Mixed Models Analysis — The apriori threshold for significance was a= 0.05. The p value reflects the test of an interaction between condition and intervention period (days 7-14, squared)

5. Secondary Outcome: Attention Network Task (ANT)
Description: Behavioural measure of general attentional control, using reaction time. A larger number suggests lower attention control, whereas a smaller number suggests greater attention control.
Time Frame: as for outcome 1
Population: Participants were only included on this analyses if they had data for all time points. 10 participants were not included (2 from ATT, 8 from control).
Measure: Mean (Standard Deviation); unit: miliseconds
Arm/Group | Attention Training Technique | Control Condition
Number analyzed (Participants) | 32 | 36
miliseconds
  Visit 1 | 104.60 (40.74) | 108.82 (40.59)
  Visit 2 | 80.02 (33.43) | 85.58 (31.85)
  Visit 3 | 80.51 (44.14) | 76.76 (42.10)
Statistical Analysis 1: Comparison: Attention Training Technique vs Control Condition; Test type: Superiority; p = .46, ANOVA — [p-value comment as in outcome 3, analysis 1]

6. Secondary Outcome: Metacognition Questionnaire 30 (MCQ-30) Cognitive Self Consciousness Subscale
Description: Self-report measure of focus of attention. Scores range from 6- 24. Greater scores represent greater self-focused attention.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Attention Training Technique | Control Condition
Number analyzed (Participants) | 34 | 44
score on a scale
  Visit 1 | 17.21 (3.41) | 17.84 (3.88)
  Visit 2 | 17.56 (3.27) | 18.02 (4.07)
  Visit 3 | 16.65 (3.56) | 17.82 (4.31)
Statistical Analysis 1: Comparison: Attention Training Technique vs Control Condition; Test type: Superiority; p = .53, ANOVA — [p-value comment as in outcome 3, analysis 1]

7. Secondary Outcome: Metacognitions Questionnaire 30 (MCQ-30) Negative Beliefs About the Uncontrollability of Thoughts and Danger Subscale
Description: Self-report measure of beliefs about the uncontrollability and dangerousness of worry. Scores range from 6-24. Greater scores represent greater negative beliefs about worry.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Attention Training Technique | Control Condition
Number analyzed (Participants) | 34 | 44
score on a scale
  Visit 1 | 17.68 (3.65) | 18.07 (3.59)
  Visit 2 | 17.00 (3.68) | 17.84 (3.77)
  Visit 3 | 15.21 (4.30) | 17.36 (3.62)
Statistical Analysis 1: Comparison: Attention Training Technique vs Control Condition; Test type: Superiority; p = .07, ANOVA — [p-value comment as in outcome 1, analysis 1]

8. Secondary Outcome: Attention Control Scale
Description: Self-report measure of attentional control. Scores range from 20-80. Greater scores indicate greater self-reported attention control.
Time Frame: as for outcome 1
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Attention Training Technique | Control Condition
Number analyzed (Participants) | 34 | 43
score on a scale
  Visit 1 | 47.59 (9.78) | 44.09 (7.68)
  Visit 2 | 46.62 (8.21) | 44.61 (7.28)
  Visit 3 | 49.17 (10.62) | 46.72 (8.31)
Statistical Analysis 1: Comparison: Attention Training Technique vs Control Condition; Test type: Superiority; p = .58, ANOVA — the apriori threshold for significance was 0.05 The p value reflects the test of an interaction between condition and time

9. Secondary Outcome: Dot Probe
Description: Behavioural measure of attentional bias to threat related words, measured in reaction time. A larger positive number indicates a greater bias to threat information while a negative number indicates the participant was faster to respond to neutral information.
Time Frame: as for outcome 1
Population: Participants were only included on this analyses if they had data for all time points. 17 participants were not included (10 from ATT, 7 from control). A substantial amount of data was lost due to a technical issue with the computer.
Measure: Mean (Standard Deviation); unit: miliseconds
Arm/Group | Attention Training Technique | Control Condition
Number analyzed (Participants) | 24 | 37
miliseconds
  Visit 1 | 6.78 (19.12) | -1.75 (19.54)
  Visit 2 | 2.14 (15.85) | -2.42 (19.66)
  Visit 3 | 0.65 (17.81) | -5.83 (23.37)
Statistical Analysis 1: Comparison: Attention Training Technique vs Control Condition; Test type: Superiority; p = .86, ANOVA — [p-value comment as in outcome 3, analysis 1]

10. Secondary Outcome: Southampton Mindfulness Questionnaire
Description: Self-report measure of mindfulness. Scores range from 0-96. Greater scores indicate greater self-reported mindfulness.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Attention Training Technique | Control Condition
Number analyzed (Participants) | 34 | 44
score on a scale
  Visit 1 | 36.09 (12.93) | 32.21 (11.93)
  Visit 2 | 36.38 (13.41) | 34.77 (12.21)
  Visit 3 | 43.88 (12.47) | 38.68 (13.35)
Statistical Analysis 1: Comparison: Attention Training Technique vs Control Condition; Test type: Superiority; p = .39, ANOVA — [p-value comment as in outcome 3, analysis 1]

11. Other Pre Specified Outcome: UPPS-P
Description: Self-report measure of impulsivity. Scores range from 12 to 48. Greater scores indicate greater negative urgency.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Attention Training Technique | Control Condition
Number analyzed (Participants) | 34 | 44
score on a scale
  Visit 1 | 29.85 (6.42) | 31.98 (7.12)
  Visit 2 | 28.71 (7.15) | 31.43 (7.28)
  Visit 3 | 28.32 (6.59) | 29.39 (8.28)

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Attention Training Technique | Control Condition
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/44
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/44
Other Adverse Events (participants affected / at risk) | 0/34 | 0/44

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-10): https://cdn.clinicaltrials.gov/large-docs/82/NCT03216382/Prot_SAP_000.pdf